CLINICAL TRIAL: NCT02082275
Title: Implementation and Evaluation of the OB Nest Project at the Point of Care: Redefining Continuity of Care for Expectant Mothers.
Brief Title: OB Nest; Redefining Continuity of Care for Expectant Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Abimbola Famuyide, Associate Professor of Obstetrics-Gynecology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-009513
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy
Keywords: Prenatal Care; Obstetrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OB Nest (Experimental): OB Nest is designed to reduce the number of pre-planned visits with their OB provider and replace the in-clinic visits with a direct and constant support from an assigned nursing team. OB Nest will empower moms-to-be to take ownership of their prenatal care by providing a wealth of resources.
  Interventions: Other: OB Nest
- Traditional Prenatal care (No Intervention): Traditional prenatal visits in clinic with OB providers.

INTERVENTIONS:
Other: OB Nest — * Reduction in the number of clinic office visits
  * Assignment to a specific nursing care team
  * Support and direct interaction available through tools which supports mom's empowerment to address her concerns, care for herself and connect with OB as necessary between clinic visits.
  * Empower and enable mothers to complete at home measurements for fetal heart rate, weight, and blood pressures.
  * Augmentation of in-person visits between care providers and patients with video conversations.
  * Maternal outcomes will be monitored through surveys and questionnaires.
  Arms: OB Nest

SUMMARY:
The study defines a new model of prenatal care called OB Nest which will be compared to the traditional model of prenatal care. OB nest is intended to create an experience for patients that feels more connected and patient-centered, allowing the patient to visit the clinic less frequently while offering increased communication with the OB nurses and providers through new tools provided to the patient. The goal of the project is to promote patient-centered care through a new prenatal care program based on constant and direct support from a nursing team, meeting the on-demand needs of expecting mothers as they rise, and as thus, redesigning the need and timing of on-site appointment with providers. Pregnant women randomized to the OB Nest cohort will see the number of pre-planned visits with their providers decreased and replaced with more direct and constant support and interaction with an assigned nursing team.

DETAILED DESCRIPTION:
OB Nest is a model designed to promote increased patient-centered care during pregnancy. OB Nest care will allow for more flexibility, decrease interruptions to your productivity, while continuing to maintain safety for you and your infant. This model of care is anticipated to allow you more access to your health care team during your pregnancy.

This study will compare OB Nest, a new model of prenatal care, to the existing traditional model of prenatal care. The plan is to have about 300 low-risk mothers take part in this study. Eligible patients will be randomized to one of two groups; The Traditional Prenatal care Group or the OB Nest Group. Mothers will have an equal chance of being assigned to the OB Nest group. Mothers randomized to the OB Nest intervention will be assigned to a nursing care team comprised of one to three nurses and see their initial eleven planned appointments with their provider reduced to six. Mothers will still be able to request additional in-office visits with their provider and/or the provider require additional in-office visits to monitor mother and infants safety/care.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Documented gestational age less than 13 weeks.
* Pregnancy documented as low risk (See high risk exclusion criteria below)
* Able to read and understand English
* Able to provide informed consent (i.e. no impairments or barriers)

Exclusion Criteria:

Clinical judgment that determines that the pregnancy is at high risk for complications.

Any of the following high risk factors would disqualify the mother for the study:

* Severe hypertension (>160/110)
* Possible ectopic
* Congenital adrenal hypertension
* Prior PE/DVT/stroke
* Anticoagulation during prior pregnancy (e.g. antiphospholipid antibody syndrome)
* Prosthetic heart valve (non-bio)
* Pulmonary hypertension
* Mothers currently taking Immunosuppressants, Prednisone > 10mg per day, antipsychotic (e.g. lithium, Haldol, Zyprexa), chemotherapy
* Recurrent pregnancy loss (>2 losses)
* Current maternal malignancy
* Prior myocardial infarction/cardiomyopathy
* Bio-prosthetic heart valves
* Marfan syndrome
* Active liver disease (e.g. hepatitis)
* Congenital heart disease
* Coagulopathies including thrombophilias and bleeding disorders.
* Pre-existing diabetes
* Genetic disease/CF testing/anomalies in prior child
* Incompetent cervix (prior cerclage)
* Triplets or quads diagnosed by REI or ultrasound.
* Isoimmunization (Rh, Kell, etc.)
* History of transplant or currently on Dialysis
* Recurrent pregnancy loss (antiphospholipid antibody syndrome or collagen vascular disease)
* Chronic hypertension
* Prior 2nd or 3rd trimester loss
* HIV
* Inflammatory bowel disease
* Asthma and currently on steroid to control disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Expectant mothers satisfaction of prenatal care | 36 weeks
  At 36 weeks the expectant mother will complete a survey that assessed their satisfaction of the prenatal care received using a validated scale.

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola Famuyide, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Theiler RN, Butler-Tobah Y, Hathcock MA, Famuyide A. OB Nest randomized controlled trial: a cost comparison of reduced visit compared to traditional prenatal care. BMC Pregnancy Childbirth. 2021 Jan 21;21(1):71. doi: 10.1186/s12884-021-03557-3. PMID 33478433
- [Derived] Butler Tobah YS, LeBlanc A, Branda ME, Inselman JW, Morris MA, Ridgeway JL, Finnie DM, Theiler R, Torbenson VE, Brodrick EM, Meylor de Mooij M, Gostout B, Famuyide A. Randomized comparison of a reduced-visit prenatal care model enhanced with remote monitoring. Am J Obstet Gynecol. 2019 Dec;221(6):638.e1-638.e8. doi: 10.1016/j.ajog.2019.06.034. Epub 2019 Jun 19. PMID 31228414
- [Derived] Ridgeway JL, LeBlanc A, Branda M, Harms RW, Morris MA, Nesbitt K, Gostout BS, Barkey LM, Sobolewski SM, Brodrick E, Inselman J, Baron A, Sivly A, Baker M, Finnie D, Chaudhry R, Famuyide AO. Implementation of a new prenatal care model to reduce office visits and increase connectivity and continuity of care: protocol for a mixed-methods study. BMC Pregnancy Childbirth. 2015 Dec 2;15:323. doi: 10.1186/s12884-015-0762-2. PMID 26631000